CLINICAL TRIAL: NCT03192306
Title: A Multicenter, Placebo-Controlled, Randomized, Double-Blind Study of the Safety and Efficacy of Merlin (Ethanol and Glycolic Acid Mixture) for the Episodic Treatment of Recurrent Herpes Labialis
Brief Title: Safety and Efficacy of Merlin (Ethanol and Glycolic Acid Mixture) for Episodic Treatment of Cold Sores
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Topical Remedy (Industry)
Collaborators: Benu BioPharma, LLC (Industry); Accelovance (Industry); Optimal Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TR-H-212
Record Dates: First submitted 2017-06-13; First posted 2017-06-20 (Actual); Results first posted 2018-08-16 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Recurrent Herpes Labialis
Keywords: Herpes Labialis; Cold Sore
MeSH Terms: conditions — Herpes Labialis | interventions — Neurofibromin 2; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Merlin (Active Comparator): glycolic acid and ethanol mixture
  Interventions: Drug: Merlin
- Ethanol (Placebo Comparator)
  Interventions: Drug: Ethanol

INTERVENTIONS:
Drug: Merlin — glycolic acid/ethanol solution
  Arms: Merlin
Drug: Ethanol — Ethanol solution
  Arms: Ethanol

SUMMARY:
The purpose of this study is to determine if Merlin, a mixture of ethanol and glycolic acid, is safe and effective in the treatment of cold sores.

Subjects who meet the requirements to participate in the study will be put randomly, and equally, into one of two groups: 1) a group receiving Merlin to treat their cold sore; or 2)a group receiving a placebo of just ethanol to treat their cold sore. Neither the subject nor the site will know which treatment they will be getting. Once the subject has been assigned to a treatment group, they will be given a kit containing a bottle of the treatment and special swabs to apply the liquid. The subject will be told to take the kit home and wait until they think they are starting to get a cold sore.

Once a subject begins to see something that they think is the start of a cold sore, they are to immediately call the clinic. Once the clinic confirms that the subject is in fact starting to get a cold sore, the subject will be told to open the kit and begin treatment. From the start of treatment, there will be twelve (12) treatments, with either Merlin or placebo, applied six (6) hours apart, up to 3 per day, over the next 96 hours (4 days). Each treatment of Merlin or placebo is made up of three (3) applications given twenty (20) minutes apart, for a total of thirty-six (36) applications. For each application, the subject will use the special swab to put the Merlin or placebo solution on their cold sore.

Subjects will need to report daily to the clinic for a minimum of 3 consecutive days, until either the cold sore is completely healed or 14 days from the start of treatment, whichever comes first. At each clinic visit the cold sore will be observed to determine at what stage it is at or if it has healed. The subject will also be asked how they are feeling.

Subjects will also be told to record in a diary the time of each application of Merlin or placebo. They will also be asked to record the stage of their lesion and how much pain, if any, related to the cold sore, that they are feeling.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject 18-75 years of age
* Female subjects must be using a medically acceptable form of birth control during the study. Acceptable birth control measures include, but are not limited to: abstinence, oral contraceptive pills or patch, injectable contraception, barrier contraceptives (condom, diaphragm with spermicide), IUD, vaginal contraceptive ring, surgical (hysterectomy, tubal ligation), vasectomized partner, and natural post-menopausal inability to conceive. Menopause is defined for this protocol as starting one year after the time of the last menstrual period.
* Subject must have a history of recurrent herpes labialis and report at least 3 separate recurrences (i.e. multiple herpetic lesions in one outbreak count as only one episode) during the preceding 12 months.
* Subject must have a history of experiencing prodromal symptoms of cold sores (e.g. itching, tingling, or burning) during at least half of their previous cold sore episodes.
* Subject must have a history of at least half of their cold sore episodes producing classical lesions (i.e., episodes that progressed through macule, papule, vesicle, crust, and healed).
* Subject must provide voluntary written informed consent to participate in this study.
* Subject is able to appear for a clinic visit within 24 hours from the time of treating cold sore and is able to return to the clinic for the full 14 day duration of the study if necessary.

Exclusion Criteria:

* Subjects with evidence of active malignancy or immunodeficiency disease within the last 30 days. Subjects who have completed therapy and are considered unlikely to relapse or who have had surgery and do not have any evidence of disease, are eligible for the study.
* Subject requires chronic use of immunomodifying drugs (e.g. systemic steroids) or topical steroids on or near the face; use of inhaled steroids does not exclude a subject from the study. If a subject is unlikely to get through the Treatment Phase of the protocol without requiring the use of an immunomodifying drug for a chronic condition the subject should be excluded.
* Subject requires chronic use of anti-viral medication. In females of childbearing potential, a positive urine pregnancy test at time of screening.

Nursing mothers.

* Subject has abnormal skin conditions (e.g. acne, eczema, rosacea, psoriasis, albinism, or chronic vesiculobullous disorders) that occur in the area ordinarily affected by cold sores or has significant facial hair in the area of the cold sore that might affect the normal course of the cold sore or might impair accurate evaluation of the cold sore lesion.
* Subject has had a vaccine for herpes simplex virus type 1 (typically oral herpes) or 2 (typically genital herpes).
* Subject is currently enrolled in another clinical trial involving the use of a drug and/or a device.
* Subject requires chronic use of analgesics or non-steroidal anti-inflammatory agents (NSAIDs) except for low doses of aspirin (less than 325 mg/day) used for cardiovascular purposes. If a subject is unlikely to get through the Treatment Phase of the protocol without requiring the use of analgesia for a chronic condition, e.g. back pain, recurrent daily headaches, the subject should be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2018-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Bart, Sr., M.D., Principal Investigator — Optimal Research Rockville MD; Murray A Kimmel, DO, Principal Investigator — Optimal Research Melbourne FL; Daniel H Brune, MD, Principal Investigator — Optimal Research Peoria IL; Stephen Daniels, DO, Principal Investigator — Optimal Research Austin TX; Randle T Middleton, MD, Principal Investigator — Optimal Research Huntsville AL; Patrick Yassini, MD, Principal Investigator — Optimal Research San Diego CA
Locations (6):
- United States (6):
  - Optimal Research, Huntsville, Alabama
  - Optimal Research, San Diego, California
  - Optimal Research, Melbourne, Florida
  - Optimal Research, Peoria, Illinois
  - Optimal Research, Rockville, Maryland
  - Optimal Research, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Merlin | Ethanol
Started | 227 | 224
Modified Intent to Treat (MITT) (MITT represents data collected from enrolled subjects who developed a cold sore and treated.) | 76 | 80
Completed | 75 | 79
Not Completed | 152 | 145
Not completed — Did not treat cold sore during study | 149 | 143
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Participants are all those subjects enrolled and given a Treatment Kit. Only subjects who actually developed a treatable cold sore lesion were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Merlin | Ethanol | Total
Number analyzed (Participants) | 227 | 224 | 451
Age, Categorical [Count of Participants; unit: Participants] — Population: Only subjects who developed a cold sore and treated during the course of the study were analyzed.
  Participants
    number analyzed (Participants) | 76 | 80 | 156
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 73 | 77 | 150
    >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Only those subjects who developed a cold sore and treated were analyzed.
  Years
    number analyzed (Participants) | 76 | 80 | 156
    (all) | 41.4 (11.84) | 42.7 (12.8) | 42.1 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only subjects who had a cold sore and treated during the course of the study were summarized in demographics tables
  Participants
    number analyzed (Participants) | 76 | 80 | 156
    Female | 56 | 62 | 118
    Male | 20 | 18 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only subjects who developed a cold sore and treated during the course of the study were analyzed.
  Participants
    number analyzed (Participants) | 76 | 80 | 156
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 5 | 5 | 10
    White | 68 | 66 | 134
    More than one race | 2 | 3 | 5
    Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Number; unit: participants] — Population: Only subjects who developed a cold sore lesion and treated were analyzed.
  participants
    United States: number analyzed (Participants) | 76 | 80 | 156
    United States | 76 | 80 | 156

OUTCOME MEASURES:

1. Primary Outcome: Clinician Assessed Duration of the Classical Herpetic Lesion
Description: The time in hours from beginning of treatment to onset of Stage 6 (residual swelling) or Stage 7 (complete healing) if Stage 6 never observed
Time Frame: From time of beginning of treatment until onset of Lesion Stage 6 or Stage 7, if Stage 6 never observed, with a maximum of 14 days.
Population: Only those subjects who developed a classical cold sore lesion, i.e. exhibited Stages 3, 4 or 5, during the course of the trial and treated were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Merlin | Ethanol
Number analyzed (Participants) | 64 | 74
hours | 162.7 (68.4) | 163.6 (74.9)

2. Secondary Outcome: Clinician Assessed Duration of the Herpetic Episode
Description: For classical lesions: the time in hours from the beginning of the treatment until loss of hard crust (Stage 6); for non-classical lesions the time from the beginning of treatment until complete resolution of all local signs and symptoms (Stage 7)
Time Frame: For classical lesions: from the beginning of the treatment until loss of hard crust (Stage 6); for non-classical lesions the time from the beginning of treatment until complete resolution of all local signs and symptoms (Stage 7) - maximum of 14 days
Population: Subjects who developed a cold sore lesion and treated during the course of the trial. One subject in the Merlin cohort was lost to follow-up, did not complete the study and was therefore excluded from this analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Merlin | Ethanol
Number analyzed (Participants) | 75 | 80
hours | 151.1 (70.9) | 158.6 (74.5)

3. Secondary Outcome: Clinician Assessed Duration Until Complete Healing of the Herpetic Episode
Description: The time, in hours, from the beginning of treatment to onset of Stage 7
Time Frame: From the beginning of treatment to onset of Stage 7 - maximum of 14 days
Population: Subjects who developed a cold sore and treated during the course of the trial. One subject in the Merlin cohort was lost to follow-up, did not complete the study and was therefore excluded from this analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Merlin | Ethanol
Number analyzed (Participants) | 75 | 80
hours | 223.4 (83.2) | 222.0 (86.4)

4. Secondary Outcome: Clinician Assessed Prevention of Progression to Classical Lesion
Description: Proportion of subjects in each treatment group who do not display classical lesions
Time Frame: 14 days maximum
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Merlin | Ethanol
Number analyzed (Participants) | 75 | 80
Participants | 12 | 6

5. Secondary Outcome: Clinician Assessed Lesion Size
Description: Maximum lesion area for ulcerative lesions during Stages 3-5
Time Frame: 14 days maximum
Population: Subjects who developed a classical herpetic lesion during the course of the trial.
Measure: Mean (Standard Deviation); unit: square mm
Arm/Group | Merlin | Ethanol
Number analyzed (Participants) | 64 | 74
square mm | 46.8 (50.2) | 36.2 (43.7)

6. Secondary Outcome: Clinician Assessed Duration of the Herpetic Lesion Hard Scab
Description: Duration of the hard crust (Stage 5)
Time Frame: From start of Stage 5 to loss of hard crust - maximum of 14 days
Population: Only those subjects who developed a cold sore with a hard scab (Stage 5) were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Merlin | Ethanol
Number analyzed (Participants) | 74 | 80
hours | 66.6 (56.8) | 65.9 (62.3)

7. Secondary Outcome: Subject Assessed Duration of Pain
Description: Time of first occurrence of at least mild pain to consistent scoring of no pain
Time Frame: From time of first occurrence of at least mild pain to time of consistent scoring of no pain - maximum 14 days
Population: Subjects with cold sore lesions pain assessment. One subject in the Merlin cohort was lost to follow-up, did not complete the study and was therefore excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Merlin | Ethanol
Number analyzed (Participants) | 75 | 80
Participants
  First Treatment: number analyzed (Participants) | 75 | 79
  First Treatment: No Pain | 31 | 35
  First Treatment: Mild | 40 | 37
  First Treatment: Moderate | 4 | 7
  First Treatment: Severe | 0 | 0
  Second Treatment: No Pain | 33 | 32
  Second Treatment: Mild | 30 | 40
  Second Treatment: Moderate | 12 | 7
  Second Treatment: Severe | 0 | 1
  Third Treatment: No Pain | 29 | 32
  Third Treatment: Mild | 28 | 38
  Third Treatment: Moderate | 18 | 7
  Third Treatment: Severe | 0 | 3
  Fourth Treatment: number analyzed (Participants) | 73 | 78
  Fourth Treatment: No Pain | 31 | 35
  Fourth Treatment: Mild | 30 | 35
  Fourth Treatment: Moderate | 11 | 6
  Fourth Treatment: Severe | 1 | 2
  Fifth Treatment: number analyzed (Participants) | 73 | 74
  Fifth Treatment: No Pain | 33 | 34
  Fifth Treatment: Mild | 30 | 30
  Fifth Treatment: Moderate | 9 | 9
  Fifth Treatment: Severe | 1 | 1
  Sixth Treatment: number analyzed (Participants) | 72 | 70
  Sixth Treatment: No Pain | 38 | 33
  Sixth Treatment: Mild | 23 | 28
  Sixth Treatment: Moderate | 9 | 9
  Sixth Treatment: Severe | 2 | 0
  Seventh Treatment: number analyzed (Participants) | 65 | 65
  Seventh Treatment: No Pain | 38 | 31
  Seventh Treatment: Mild | 16 | 29
  Seventh Treatment: Moderate | 10 | 5
  Seventh Treatment: Severe | 1 | 0
  Eighth Treatment: number analyzed (Participants) | 59 | 59
  Eighth Treatment: No Pain | 40 | 30
  Eighth Treatment: Mild | 10 | 24
  Eighth Treatment: Moderate | 7 | 5
  Eighth Treatment: Severe | 2 | 0
  Ninth Treatment: number analyzed (Participants) | 55 | 55
  Ninth Treatment: No Pain | 38 | 31
  Ninth Treatment: Mild | 10 | 19
  Ninth Treatment: Moderate | 5 | 5
  Ninth Treatment: Severe | 2 | 0
  Tenth Treatment: number analyzed (Participants) | 51 | 51
  Tenth Treatment: No Pain | 32 | 26
  Tenth Treatment: Mild | 11 | 22
  Tenth Treatment: Moderate | 5 | 3
  Tenth Treatment: Severe | 3 | 0
  Eleventh Treatment: number analyzed (Participants) | 47 | 52
  Eleventh Treatment: No Pain | 32 | 31
  Eleventh Treatment: Mild | 9 | 16
  Eleventh Treatment: Moderate | 4 | 5
  Eleventh Treatment: Severe | 2 | 0
  Twelfth Treatment: number analyzed (Participants) | 45 | 51
  Twelfth Treatment: No Pain | 33 | 32
  Twelfth Treatment: Mild | 9 | 15
  Twelfth Treatment: Moderate | 2 | 4
  Twelfth Treatment: Severe | 1 | 0
  Max Severity Post Treatment: number analyzed (Participants) | 70 | 78
  Max Severity Post Treatment: No Pain | 45 | 47
  Max Severity Post Treatment: Mild | 14 | 20
  Max Severity Post Treatment: Moderate | 9 | 8
  Max Severity Post Treatment: Severe | 2 | 3

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the course of treatment until the herpetic lesion healed, or for 14 days from the first report of a cold sore, whichever occurred first, for all those who developed a cold sore in the study, and for two weeks after completion of treatment or for two weeks after the 14 day Treatment Phase study period.
Arm/Group | Merlin | Ethanol
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/80
Other Adverse Events (participants affected / at risk) | 10/76 | 4/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Merlin (N=76) | Ethanol (N=80)
Diahrrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Seborrhoeic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any manuscript, abstract, or other publication or presentation of results or information arising in connection with the study must be prepared in conjunction with Topical Remedy, LLC.

DOCUMENTS (2):
  • Study Protocol (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT03192306/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT03192306/SAP_001.pdf